CLINICAL TRIAL: NCT01911117
Title: Evaluating the Correction of Non-invasive Estimated Continuous Cardiac Output in Cardiac Surgical Patients
Status: Withdrawn | Type: Observational
Why Stopped: No man power
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Yen Chin Liu, Visiting Staff, Department of Anesthesiology Chief, National Cheng-Kung University Hospital
Other Study IDs: A-ER-102-080
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiac Surgical Patients: Patients who undergo cardiac surgery will be included in this study.
  1. Patients undergo cardiac surgery and are over 18 years of age.
  2. Patients need bypass machine for their cardiac surgery and traditional CO measurement.
  3. Patients who are competent to understand the study and provide written informed consent and participate in outcome measurements.

SUMMARY:
In one previous study, esCCO was compared with continuous thermodilution CO (TDCO), measurements in 36 postoperative cardiac surgery patients, showing a bias (mean difference) of -0.06 and a precision (1 SD) of 0.82 L/min. In addition, esCCO was compared with intermittent bolus TDCO, showing a correlation coefficient of 0.82 (P < 0.001, n = 24), a bias of -0.63, and a precision of 1.01 L/min (n = 119). The results of clinical use of esCCO suggest that its measurement accuracy is comparable to the thermodilution method in general population. However, no any intraoperative comparison for cardiac surgery patients was reported before. This study is designed for the accuracy in the patients undergoing cardiac surgery.

Specific aims:

1. To investigate the correlation of esCCO and the traditional CO measurement in cardiac surgical patients.
2. To investigate the intraoperative t accuracy of time point between ecCCO and traditional CO measurement for patients undergoing bypass cardiac surgery.

DETAILED DESCRIPTION:
Determination of cardiac output (CO) is often desirable for assessing a patient's hemodynamic condition during the surgery requiring cardiopulmonary bypass. However, the current methods of continuous CO measurement are still based on invasive technique, such as thermodilution via pulmonary artery catheter (Swan-Ganz), transpulmonary thermodilution via PiCCO kit, or pulse contour analysis via arterial line (FloTrac or PiCCO). Noninvasive CO measurement to all patients is currently impractical, because most measurement methods available are based on invasive techniques. However, two developing trends for this kind of monitor had occurred. There are one shifting toward noninvasive technologies and the other trend toward continuous measurement rather than intermittent measurement. Therefore, continuous CO (CCO) monitoring with less invasive would be desirable.

The pulse contour method is one of the technologies used for min-invasive monitoring of CO. It is based on the relationship between arterial blood pressure and stroke volume and has been greatly improved since early 1950s. Arterial waveform-based CO is frequently used in current medical practice, but it still requires arterial puncture. Pulse wave transit time has been proven to have good correlation with stroke volume. Pulse wave transit time consists of a pre-ejection period, pulse wave transit time through the artery, and pulse wave transit time through the peripheral arteries, which compensates for the effect of changes in systemic vascular resistance (SVR). Based on the relationship between pulse wave transit time and stroke volume, the noninvasive device, estimated CCO (esCCO), via measuring electrocardiogram (ECG), pulse oximeter wave, and arterial blood pressure had been developed by Sugo et al.. It has the great advantage to simplify CO measurement by combining the results of these familiar noninvasive monitoring techniques. Thus, it may be a useful technique for optimizing medical treatment.

In one previous study, esCCO was compared with continuous thermodilution CO (TDCO), measurements in 36 postoperative cardiac surgery patients, showing a bias (mean difference) of -0.06 and a precision (1 SD) of 0.82 L/min. In addition, esCCO was compared with intermittent bolus TDCO, showing a correlation coefficient of 0.82 (P < 0.001, n = 24), a bias of -0.63, and a precision of 1.01 L/min (n = 119). The results of clinical use of esCCO suggest that its measurement accuracy is comparable to the thermodilution method in general population. However, no any intraoperative comparison for cardiac surgery patients was reported before. This study is designed for the accuracy in the patients undergoing cardiac surgery.

Specific aims

1. To investigate the correlation of esCCO and the traditional CO measurement in cardiac surgical patients.
2. To investigate the intraoperative t accuracy of time point between ecCCO and traditional CO measurement for patients undergoing bypass cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergo cardiac surgery and are over 18 years of age.
2. Patients need bypass machine for their cardiac surgery and traditional CO measurement.
3. Patients who are competent to understand the study and provide written informed consent and participate in outcome measurements.

Exclusion Criteria:

* Patients are over 75 years of age. Patients are unable to read or write the informed consent, any condition that could interfere with the interpretation of outcome assessments, pregnant or lactating women. Patient with marked arrhythmias, those preoperatively receiving treatment with intra-aortic balloon bump (IABP) will also not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo cardiac surgery will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The correlation of esCCO and the traditional CO measurement in cardiac surgical patients. | 18 months
  1. Comparison Between esCCO and Thermodilution Measurements of CO for cardiac surgical patients.
  2. Check the accuracy of esCCO in cardiac surgical patients. It should be well correlated before bypass but will be inaccurate when partial bypass once start. When bypass procedure start to rewarm, it will be accurate initially but gradually well correlated within temperature corrected or heart function become normal again.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Chin Liu, Doctor, Study Chair — Department of Anesthesiology, National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Shengli Rd, Taiwan